CLINICAL TRIAL: NCT02070445
Title: Ventilation During Cardiopulmonary Bypass (CPB) for Cardiac Surgery - Effect on Pulmonary Atelectasis Post-operatively, a Pilot Study
Brief Title: Ventilation During Cardiopulmonary Bypass (CPB) for Cardiac Surgery
Status: Withdrawn | Type: Observational
Why Stopped: One of the investigators left the institution.
Sponsor: McMaster University (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Other Study IDs: 13-859
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Last update posted 2019-08-08 (Actual); Status verified 2019-03

CONDITIONS: Pulmonary Atelectasis
Keywords: CABG; pilot; ultrasound; perioperative; low tidal volume ventilation
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing CABG: Patients will have no ventilation during CABG. There will be non-invasive assessments of the lung using ultrasound at different times during the perioperative period.The first assessment will be conducted before anesthesia induction (i.e. patients will be awake). A second assessment will be conducted after anesthesiology induction, but before the beginning of surgery. A third assessment will be conducted at the end of the surgery in the operating room. And two subsequent assessments will be conducted in ICU before and after extubation.

SUMMARY:
During most types of heart surgery cardiopulmonary bypass (CPB) is used. CPB enables blood to be directed away from the heart and the lungs and pumped through the body while the heart is not beating. Surgery on the heart easier when it is not beating and bloodless area. Generally during CPB the lungs do not need to be ventilated, as no blood is flowing through the lungs and the body received oxygen from a machine (oxygenator) attached to the CPB pump.

In this study we are investigating the difference in lung collapse after heart surgery in patient who did have their lungs ventilated during CPB, compared to patients who did not have their lungs ventilated during CPB. We will use lung ultrasound scans to determine the degree of lung collapse at various time periods before and after the heart surgery. We will also investigate if ventilation during CPB will affect: a.) the rate of lung infection or pneumonia after the operation b.) the time it takes for a patient to have the breathing tube removed in the intensive care unit after the operation c.) the time for a patient to be discharged home from the hospital d.) the concentration of oxygen in the blood after the operation.

DETAILED DESCRIPTION:
Objective and Hypothesis:

To determine if continued mechanical ventilation (low tidal volume ventilation) during cardiopulmonary bypass (CPB) in adult patients undergoing elective cardiac surgery will reduce the degree of pulmonary atelectasis post-operatively, when compared to controls not ventilated during CPB.

The degree of pulmonary atelectasis will be assessed and quantified using non-invasive lung ultrasound (LUS) imaging.

We will conduct a preliminary observational study (pilot study) to assess the feasibility of this study. The pilot will be conducted on 40 patients, all of whom will be non-ventilated during CPB. The specific feasibility questions we would like to determine are: 1) the degree of atelectasis that can be demonstrated by LUS on patients that are not ventilated while on CPB, 2) the time needed to complete a LUS in the operating room (OR) and in the intensive care unit (ICU) and whether this will be efficient and possible given the busy operating room schedule, 3) to help determine the optimal time to scan patients to show the maximal degree of atelectasis, and 4) to help estimate the number of patients we will need to show a difference in atelectasis in the definitive study.

Primary hypothesis: low tidal volume ventilation during CPB for adult cardiac surgery reduces the amount of pulmonary atelectasis compared to controls not ventilated during CPB.

Background:

Respiratory dysfunction after cardiac surgery is relatively common, with an incidence anywhere from 2- 25% quoted in the literature. Pulmonary complications are a significant factor in morbidity and mortality of post-surgical patients, and therefore a burden on healthcare resources.(1)

The etiology of post CPB pulmonary dysfunction is multi-factorial, including CPB-induced systemic inflammatory response, hypothermia, surgery, anesthesia, ventilation and transfusion. (2-3) Modifications in the above-mentioned factors, amongst others, may lead to better lung function postoperatively. Strategies include reducing CPB time, or minimizing the extracorporeal surface area with the use of miniaturized circuits. The partial restoration of pulmonary artery perfusion during CPB possibly contributes to prevent pulmonary ischemia and lung dysfunction. The use of ultrafiltration to scavenge pro-inflammatory factors may be protective for lung function. (4) Similarly, the use of corticosteroids and leukocyte depletion filters may be protective. (5-6) Reducing the use of the cardiotomy suction device, as well as the contact-time between free blood and pericardium, may prove beneficial. The evidence for outcome benefit for most of these interventions is, however, weak. (3-7)

In standard care, lungs are unventilated and deflated and blood circulation is shunted away from the pulmonary vasculature during CPB. Restoration of normal perfusion results in the release of oxygen free radicals, causing lipid peroxidation with pulmonary endothelial damage (ischemia-reperfusion injury). (8-9)

Continued ventilation during CPB has been experimentally shown to preserve pulmonary arterial endothelial function. (10) A significant consequence of reperfusion injury is dysfunction of the pulmonary vascular endothelium with diminished nitric oxide (NO) production, causing secondary vasoconstriction and increased vascular permeability. This leads to pulmonary hypertension, pulmonary edema and hypoxia. (10)

Non-ventilation may result in ischemic lung injury. During bypass there is no blood flow through the pulmonary arteries. The only vascular and hence oxygen supply to the lungs is via the bronchial circulation. (11) In an experimental porcine bypass model it has been shown that bronchial artery flow is significantly decreased during CPB. (12-13) It is hypothesized that the repetitive inflation and deflation of lungs at physiological intra-alveolar pressure is necessary for normal bronchial arterial flow secondary to the cyclical compression and relaxation of the vessels. In that case, cessation of ventilation during bypass would reduce bronchial flow and predispose to ischemic lung injury. (13)

John et al (11) showed in their randomized study that ventilation during CPB with tidal volumes of 5 ml/Kg resulted in significant smaller extra-vascular lung water (measured using the Pulse Contour Cardiac Output (PiCCO) system) and a shorter time-to-extubation. However, the evidence for clear clinical benefits of maintaining ventilation during CPB is inconsistent. Problematic in these studies are the heterogeneous outcome endpoints and small sample sizes. (11;14)

This study aims to investigate if continued low volume ventilation during CPB would decrease the amount of pulmonary atelectasis present post-operatively in cardiac surgery patients. De-recruitment of lung volumes occurs during the period of non-ventilation on CPB. Atelectasis may lead to pulmonary complications post-operatively, if not addressed in the perioperative period with active lung recruitment and physiotherapy. Low-volume ventilation can be applied easily and safely in most patients undergoing CPB without hampering the surgical progress.

Lung ultrasound (LUS) will be used to grade the pulmonary atelectasis present at various points in time (both pre-operatively and during the post-operative course). LUS is a non-invasive, easy-to-use, point-of-care investigatory tool. LUS is well validated and used in the operating room and the intensive care unit to diagnosis pulmonary pathology. It has been shown to be more accurate than plain film chest X-ray in determining pulmonary consolidation, as well as other pulmonary pathology. (13) LUS has also shown tight correlation in previous studies with pulmonary CT finding. In 2012 the first International evidence-based recommendations for point-of-care LUS were published. (16) It has become a useful and widely used modality in clinical practice. (17-18)

Several ultrasound studies based on the examination of the left lower lobe during transesophageal echocardiography have confirmed the feasibility of assessing lung recruitment (19-20). Another study has shown that resolution of ventilator-associated pneumonia with antimicrobial therapy can be accurately assessed by LUS: a tight correlation was found between an increase in computed tomography (CT) lung aeration after 7-day antibiotic administration and an ultrasound re-aeration score based on observed changes in ultrasound patterns (21). Therefore, it is reasonable to hypothesize that a change in lung aeration resulting from any therapy (for example, ventilation during CPB) will be detected by corresponding changes in LUS patterns.

ELIGIBILITY:
Inclusion Criteria:

* Adult elective coronary artery bypass surgery requiring CPB

Exclusion Criteria:

* Cardiac surgery without CPB
* Complex cardiac surgery (valve repairs, combined bypass and valve repairs etc.)
* Emergency cardiac surgery
* Fibrotic lung disease
* Previous lung volume reduction surgery (CXR will be assessed pre-operatively)
* Massive blood product transfusion intra- and/or post-operatively will exclude patient
* Patients enrolled in other studies eg. SIRS study (steroid use)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Same Day Surgery Clinic
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Time to complete study in operating room and ICU | 3 months
  To assess feasibility of LUS investigation in pre-operative and post-operative patients (time required to complete study in operating room and ICU, practicality of performing LUS in a busy environment). The LUS investigations are reported to be a fast and reliable investigation. However, few data are available about its use in a perioperative setting.

SECONDARY OUTCOMES:
Assess the evolution of LUS | 3 months
  To assess the evolution of LUS during the perioperative period. Anesthesiology induction and mechanical ventilation are recognized to induce modifications in lung ventilation and aeration. Despite this, it is unclear that LUS will be able to detect these variations. Further, the optimal timing to evaluate the LUS is not known. The optimal time for LUS assessment measurement needs to take into consideration lung ventilation parameters and also practical realization in the operating room.
Determine sample size for future Randomized Control Trial | 3 months
  To allow us to determine sample size for future randomized controlled trials. As a matter of fact, the distribution of this parameter (LUS) is not well described for perioperative patients. In order to evaluate the potential effect of lung ventilation during CPB, we first need to get an accurate estimation of LUS in the control (unventilated) population. This data will allow us to clearly define the hypothesis to test with regard to the expected treatment effect of lung ventilation during CPB.

CONTACTS AND LOCATIONS:
Overall Officials: Summer Syed, MD, Principal Investigator — McMaster University and Hamilton Health Sciences
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Taggart DP, el-Fiky M, Carter R, Bowman A, Wheatley DJ. Respiratory dysfunction after uncomplicated cardiopulmonary bypass. Ann Thorac Surg. 1993 Nov;56(5):1123-8. doi: 10.1016/0003-4975(95)90029-2. PMID 8239811
- [Background] Apostolakis EE, Koletsis EN, Baikoussis NG, Siminelakis SN, Papadopoulos GS. Strategies to prevent intraoperative lung injury during cardiopulmonary bypass. J Cardiothorac Surg. 2010 Jan 11;5:1. doi: 10.1186/1749-8090-5-1. PMID 20064238
- [Background] Asimakopoulos G, Smith PL, Ratnatunga CP, Taylor KM. Lung injury and acute respiratory distress syndrome after cardiopulmonary bypass. Ann Thorac Surg. 1999 Sep;68(3):1107-15. doi: 10.1016/s0003-4975(99)00781-x. PMID 10510030